CLINICAL TRIAL: NCT02697045
Title: Nautralsitic, Open-label, Single Arm Study Evaluating Effects of Aripiprazole LAI on Phychosocial&Congitive Functioning, Patient Reported Acceptability of Treatment Regarding QoL, Subjective Well-being Under Neuroleptic Medication in Sch
Brief Title: Effects of Aripiprazole (LAI) on Phychosocial/Cognitive Functioning, pt Reported AcceptabilityofTreatment in Sch
Acronym: ARILAI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Abdi İbrahim Otsuka (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 031-409-00036
Record Dates: First submitted 2016-02-23; First posted 2016-03-03 (Estimated); Last update posted 2019-03-06 (Actual); Status verified 2019-03

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Quality of Life; Functionality; Long Acting Injectable; Aripiprazole; Naturalistic; Open-label; Single Arm; Uncontrolled Study
MeSH Terms: conditions — Schizophrenia | interventions — Aripiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ARIPIPRAZOLE (Other): ABILIFY MAINTENA 400 MG LAI Aripiprazole 400mg, IM, Once a month
  Interventions: Drug: Aripiprazole 400mg LAI

INTERVENTIONS:
Drug: Aripiprazole 400mg LAI — Aripiprazole 400mg, IM, Once a month
  Other Names: ABILIFY

SUMMARY:
Nautralsitic, Open-label, Single Arm, Uncontrolled Study Evaluating the Effects of Long Acting Injectable (LAI) on Phychosocial Functioning Congitive Functioning and Patient Reported Acceptability of Treatment 'Reported Acceptability of Treatment' Regarding Quality of Life Subjective Well-being Under Neuroleptic Medication in Schizophrenia Patients

DETAILED DESCRIPTION:
Primary Objective

* To evaluate the efficacy of aripiprazole long acting injectable form in Turkish patients with schizophrenia on psychosocial functioning, quality of life and patient reported acceptability of treatment. Secondary Objective(s)
* To evaluate the cognitive functioning of the patients
* To evaluate positive and negative symptoms of the Aripiprazole Long Acting Injectable (LAI),
* To evaluate adherence of Aripiprazole Long Acting Injectable (LAI) treatment,
* To evaluate tolerability of Aripiprazole Long Acting Injectable (LAI).

ELIGIBILITY:
* Inclusion Criteria:

  * Participants 18-45 of years age fulfilling DSM-IV-TR diagnostic criteria of schizophrenia,
  * Disease history of ≤ 3 years (≤ 3 years after the emergence of first psychotic symptoms),
  * A history of symptom exacerbation or relapse when not receiving antipsychotics therefore requiring maintenance antipsychotic treatment,
  * Informed written consent,
  * Not on any antipsychotic treatment at least for 3 months or requiring a switch in treatment for any reason (lack of efficacy/ inadequate response to current antipsychotic(s), intolerance, nonadherence), and with the potential to benefit from extended treatment with an LAI formulation, in the investigator's opinion.
  * Lack of efficacy is defined as subjects with a baseline total PANSS score ≥70 or ≥2 items scoring ≥4 in the Positive or Negative Symptom Subscale
  * Lack of tolerability is defined as the presence of clinically relevant side effects with the previous antipsychotic medication.
  * Being literate in order to be able to answer the self report scales.
* Exclusion Criteria:

  * DSM-IV-TR diagnosis other than schizophrenia or experiencing acute depressive symptoms in the past 30 days requiring ADT depending on the clinical decision of the investigator.
  * Antipsychotic resistant or refractory schizophrenia
  * A history of failure to clozapine treatment or response to clozapine treatment only.
  * Significant risk of violent behavior or risk of self-harm
  * Currently meets DSM-IV-TR criteria for alcohol and substance dependence
  * Any clinically significant medical or neurological disorder
  * Any medically significant abnormal laboratory test or ECG result at screening
  * Pregnant, lactating.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2017-01-04 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy of aripiprazole long acting injectable form in Turkish patients with schizophrenia on psychosocial functioning assesed with psychosocial functioning scale | 24 weeks
To evaluate the efficacy of aripiprazole long acting injectable form in Turkish patients with schizophrenia quality of life assesed with Heinrich's quality of life scale | 24 weeks
To evaluate the efficacy of aripiprazole long acting injectable form in Turkish patients with schizophrenia patient reported acceptability of treatment assesed with Subjective Well Being Under Neuroleptic Treatment Scale | 24 weeks

SECONDARY OUTCOMES:
To evaluate the cognitive functioning of the patients assesed with PANNS Cognitive Items | 24 weeks
To evaluate positive and negative symptoms of the Aripiprazole Long Acting Injectable (LAI), | 24 weeks
To evaluate adherence of Aripiprazole Long Acting Injectable (LAI) treatment, | 24 weeks
To evaluate tolerability of Aripiprazole Long Acting Injectable (LAI) | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Koksal Alptekin, Prof. Dr, Principal Investigator — Dokuz Eylul Universitesi Psiyatri Anabilim Dalı
Locations (15):
- Turkey (Türkiye) (15):
  - Çukurova Üniversitesi Tıp Fakültesi Balcalı Hastanesi Dahili Tıp Bilimleri Ruh Sağlığı ve Hastalıkları Anabilim Dalı, 01330 Balcalı/, Adana
  - Ankara Atatürk Eğitim Araştırma Hastanesi Psikiyatri Kliniği, Üniversiteler Mahallesi Bilkent Caddesi No:1 ÇANKAYA / ANKARA, Ankara
  - Ankara Üniversitesi Tıp Fakültesi Ruh Sağlığı ve Hastalıkları Anabilim Dalı, Cebeci Yerleşkesi, Cebeci Ankara, Ankara
  - Hacettepe Üniversitesi Tıp Fakültesi Ruh Sağlığı ve Hastalıkları Anabilim Dalı, Hacettepe Mh. 06230 Ankara, Ankara
  - Uludağ Üniversitesi Tıp Fakültesi Hastanesi Psikiyatri ABD, Görükle Kampusu, 16059 Görükle/Nilüfer/Bursa, Bursa
  - Erenköy Ruh ve Sinir Hastalıkları EAH Psikiyatri Polikliniği E servisi (Erkek Servisi) Eğitim Sorumlusu Başhekimlik Binası Uyku Laboratuarı 3. Kat Erenköy - Kadıköy - 34736 İstanbul, Istanbul
  - Erenköy Ruh ve Sinir Hastalıkları EAH Psikiyatri Polikliniği K servisi (Kadın Servisi) 2. Kat, Sinan Ercan Cad. No:29 Kazasker - Erenköy - Kadıköy - 34736 İstanbul, Istanbul
  - İstanbul Üniversitesi İstanbul Tıp Fakültesi Psikiyatri AD, Turgut Özal Caddesi No: 118 PK. 34093 Fatih/ İstanbul, Istanbul
  - Dokuz Eylül Üniversitesi Tıp Fakültesi Dahili Tıp Bilimleri Bölümü Ruh Sağlığı Ve Hastalıkları Anabilim Dalı Mithatpaşa Cad. No 1606 İnciraltı yerleşkesi 35340 Balçova / İzmir, Izmir
  - Ege Üniversitesi Hastanesi Ruh Sağlığı ve Hastalıkları Anabilim Dalı, Kazımdirik, 35100 Bornova/İzmir, Izmir
  - Kocaeli Üniversitesi Tıp Fakültesi Araştırma ve Uygulama Hastanesi Ruh Sağlığı ve Hastalıkları Anabilim Dalı, Eski İstanbul Yolu 10. Km. Umuttepe Yerleşkesi İzmit / Kocaeli, Kocaeli
  - Sağlık Bilimleri Üniversitesi Konya Eğitim Araştırma Hastanesi, Meram, Konya, Konya
  - Manisa Ruh Sağlığı ve Hastalıkları Hastanesi Şehitler Mh. 814 Sk. No : 28 Merkez - Manisa, Manisa
  - Mersin Üniversitesi Sağlık Araştırma ve Uygulama Merkezi Hastanesi Psikiyatri Anabilim Dalı Çiftlikköy Kampüsü 33343 Yenişehir-Mersin, Mersin
  - 19 Mayıs Üniversitesi Sağlık Uygulama ve Araştırma Merkezi Ruh Sağlığı ve Hastalıkları Anabilim Dalı Atakum / SAMSUN, Samsun

IPD SHARING:
Plan to Share IPD: Yes